CLINICAL TRIAL: NCT05544097
Title: Spectral Analysis of Bowel Sounds in Preterm Babies of Less Than 32 Weeks of Amenorrhea (WA) as Predictive Factor of Enterocolitis
Acronym: BHAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI2019_843_0025
Record Dates: First submitted 2022-09-06; First posted 2022-09-16 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Bowel Sounds; Spectral Analysis; Necrotizing Enterocolitis; Preterm Babies
Keywords: bowel sounds; spectral analysis; Necrotizing Enterocolitis; preterm babies
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Recording of the bowel sounds — Recording of the bowel sounds before and after enteral feeding three times a week with an electronical stethoscope

SUMMARY:
The recording or bowels is easy and cheap. The investigators wonder if these sounds are modified in babies with high risk of necrotizing enterocolitis. In this study, the investigators suggest to record and do a spectral analysis of 30 seconds of bowel sounds in preterm babies of less than 32WA before and after enteral nutrition, every day until the end of hospitalization. A spectral analysis will be made for each record to determine frequencies of the signal. The investigators will try to determine physiological frequencies and look for modifications in pathological situations.

ELIGIBILITY:
Inclusion Criteria:

* preterm babies of less than 32WA

Exclusion Criteria:

* preterm babies of more than 32WA,
* digestive congenital malformation

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
variation of spectral analysis of bowel sounds (frequency in Hz) before and after enteral nutrition | 36 months
  establishing spectral analysis of bowel sounds

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No